CLINICAL TRIAL: NCT00952549
Title: Facial Yoga Toning Program - A Pilot Study
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator no longer at Cleveland Clinic
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FYTP
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Facial Atrophy Related to Age

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Facial Yoga Toning Program (Experimental): Patients will be instructed on 18 exercises which are intended to strengthen and tone the muscles of facial expression. DVD is provided.
  Interventions: Procedure: Facial Yoga Toning Program

INTERVENTIONS:
Procedure: Facial Yoga Toning Program — Patients will be instructed on 18 exercises which are intended to strengthen and tone the muscles of facial expression. DVD is provided.

SUMMARY:
The primary objective of this study is to determine the efficacy of a facial yoga exercise program on appearance and to measure patient satisfaction with facial yoga practice.

DETAILED DESCRIPTION:
This is a single center prospective longitudinal pilot study of 27 subjects. The study will include 20 study subjects and 7 controls. Participants in this study will be healthy subjects 18 years and older with mild to moderate facial atrophy without a history of surgical or non-surgical treatment to the area. The study subjects will perform facial yoga and apply sunscreen (Neutrogena Helioplex SPF 55) daily. The controls will apply sunscreen alone daily for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* over age 18 years

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of facial yoga toning program on aesthetic appearance | 8 weeks
  subjects will be photographed and investigator will complete Global Aesthetic Improvement Scale to document results at baseline, 2, 4, 6, and 8 weeks

SECONDARY OUTCOMES:
subject satisfaction with facial yoga toning program | 8 weeks
  subjects will complete satisfaction survey at baseline, 2, 4, 6, and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Tung, MD, Principal Investigator — The Cleveland Clinic; Wilma Bergfeld, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No